CLINICAL TRIAL: NCT02499666
Title: Evaluation of Exercise Capacity as Measured by Peak Oxygen Uptake, Before and After Percutaneous Revascularization of Chronic Total Occlusion
Brief Title: Change in Exercise Capacity as Measured by Peak Oxygen Uptake After CTO PCI
Acronym: EXERTION
Status: Terminated | Type: Observational
Why Stopped: difficulty recruiting patients
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Khaldoon Alaswad, MD, Director, Cardiac Catheterization Laboratory, Henry Ford Health System
Other Study IDs: 9608
Record Dates: First submitted 2015-07-13; First posted 2015-07-16 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease; Angina Pectoris
Keywords: Exercise Capacity; Chronic Total Occlusion
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Percutaneous Coronary Intervention; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asymptomatic: Patients with known chronic total occlusion who are undergoing percutaneous coronary intervention wtih balloon angioplasty and coronary stent placement who are currently asymptomatic (without any chest pain or anginal equivalent) but have decreased exercise capacity or are easily fatigued. Patients will also be on dual antiplatelet therapy with aspirin and a second agent such as clopidogrel.
  Interventions: Procedure: Percutaneous Coronary Intervention; Device: Coronary stent; Drug: Clopidogrel
- Symptomatic: Patients with known chronic total occlusion who are undergoing percutaneous coronary intervention with balloon angioplasty and coronary stent placement who are currently symptomatic with chest pain or anginal equivalent.. Patients will also be on dual antiplatelet therapy with aspirin and a second agent such as clopidogrel.
  Interventions: Procedure: Percutaneous Coronary Intervention; Device: Coronary stent; Drug: Clopidogrel

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — As clinically indicated, patients will have a percutaneous balloon angioplasty and stent deployment of a chronic total occlusion (i.e., an artery that has a 100% blockage for several months).
Device: Coronary stent — As clinically indicated, patients will have a coronary stent placement into their occluded coronary artery after successful balloon angioplasty
Drug: Clopidogrel — As clinically indicated, patients who are not already on dual antiplatelet therapy will be started on a second agent such as clopidogrel.
  Other Names: Plavix

SUMMARY:
The purpose of this project is to objectively assess the change (improvement) in exercise capacity in patients undergoing routine percutaneous coronary intervention (PCI) for chronic total occlusion (CTO)

DETAILED DESCRIPTION:
PURPOSE: The purpose of this project is to objectively assess the change (improvement) in exercise capacity in patients undergoing routine percutaneous coronary intervention (PCI) for chronic total occlusion (CTO)

AIMS: The primary aim of this study is to identify any improvement in exercise capacity as measured by peak oxygen uptake (VO2) and quality of life survey, for both symptomatic and asymptomatic patients (each group will be analyzed separately). 2) The secondary aim is to identify any cardiopulmonary exercise testing (CPX) predictors of exercise improvement that may then be used for selecting optimal CTO PCI candidates

RATIONALE: Chronic Total Occlusion (CTO) of a coronary vessel is defined as 100% occlusion of a coronary artery for more than 3 months. The prevalence of coronary CTO ranges from 18-34% in patients with coronary artery disease. Because of new developments in the techniques and the available technology Chronic Total Occlusion Percutaneous Coronary Intervention (CTO PCI) has been performed more frequently. The effects of successful CTO PCI on the objective findings of CPX has never been studied before. Registry and retrospective small studies have shown that successful CTO PCI decreases angina and ischemic burden, improves left ventricular function, reduces the risk of arrhythmias, increases tolerance to acute coronary syndromes, decreases the need for coronary artery by pass surgery, and improves the patient quality of life. The American College of Cardiology - American Heart Association PCI Guidelines give this procedure a Class IIa recommendation in specialized centers with expertise in CTO PCI. The ultimate goal of coronary intervention is not only improved survival and surrogate markers like left ventricular function, but improvement of quality of life. While angina is a subjective marker of quality of life, the patient's experience of angina will depend upon the degree to which the patient engages in exertion. Many patients subconsciously or consciously adjust their routine activities and exercise level to be below the threshold at which they experience angina, shortness of breath, or fatigue. The investigators therefore aim to quantify the degree to which there is any change in exercise capacity as measured by peak oxygen uptake (VO2) and a quality of life questionnaire. This information may help future patients and physicians provide prognostic information about the potential benefits of CTO PCI. Furthermore, as a secondary aim, the investigators will evaluate any CPX predictors of post PCI improvement in exercise capacity. This information may help establish algorithms for those patients who will most benefit from CTO PCI. The investigators aim to 1- objectively quantify the negative effects of coronary CTO on the CPX parameters (peak oxygen uptake), 2- demonstrate the effects of successful CTO PCI on CPX parameters especially in asymptomatic patients 3- determine the patient and procedural findings that determine improvement in CPX parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present for percutaneous intervention of chronic total occlusion who are able and willing to perform treadmill cardiopulmonary stress testing before and after the intervention

Exclusion Criteria:

* Patients who present for percutaneous intervention of chronic total occlusion who are unable or unwilling to perform treadmill cardiopulmonary stress testing before and after the intervention

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who present for evalaution of CTO-PCI (male and female, age >18 years old) will be asked to participate in the study. Patients unable to exercise for any reason will be excluded.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Exercise Capacity | Patients will be followed up until their second cardiopulmonary exercise test, which will usually be scheduled 2-12 weeks after their percutaneous coronary intervention
  Evaluate change in exercise capacity as determined by peak VO2 by comparing pre and post percutaneous intervention cardiopulmonary exercise test results

SECONDARY OUTCOMES:
Predictors of Change in Exercise Capacity | Patients will be followed up until their second cardiopulmonary exercise test, which will usually be scheduled 2-12 weeks after their percutaneous coronary intervention
  Analyze cardiopulmonary stress test data for any variables that are predictive of improvement in exercise capacity after percutaneous intervention of chronic total occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoon Alaswad, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States